CLINICAL TRIAL: NCT00101712
Title: Efficacy and Safety of Vildagliptin Compared to Placebo in Patients With Type 2 Diabetes and Mild Hyperglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2307
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Vildagliptin Placebo

INTERVENTIONS:
Drug: vildagliptin
  Other Names: LAF237
  Arms: Vildagliptin
Drug: Vildagliptin Placebo
  Arms: Placebo

SUMMARY:
This study is not being conducted in the United States. Key long-term clinical studies have shown that people with type 2 diabetes should try to achieve overall blood glucose levels as close to normal as possible. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to placebo in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar and whose blood glucose levels are close to normal.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 22-45
* Diagnosis of type 2 diabetes for at least 8 weeks

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular complications
* Significant laboratory abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Adverse event profile after 52 weeks of treatment
Patients with HbA1c <6.5% at 12 weeks
Patients with HbA1c <6.5% at 52 weeks
Change from baseline in fasting plasma glucose at 52 weeks
Coefficient of failure for HbA1c between 24 weeks and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Investigative Site, Germany
- Novartis Investigative Site, Basel, Switzerland

REFERENCES:
- [Derived] Scherbaum WA, Schweizer A, Mari A, Nilsson PM, Lalanne G, Jauffret S, Foley JE. Efficacy and tolerability of vildagliptin in drug-naive patients with type 2 diabetes and mild hyperglycaemia*. Diabetes Obes Metab. 2008 Aug;10(8):675-82. doi: 10.1111/j.1463-1326.2008.00850.x. Epub 2007 Nov 22. PMID 18248490
- [Derived] Mari A, Scherbaum WA, Nilsson PM, Lalanne G, Schweizer A, Dunning BE, Jauffret S, Foley JE. Characterization of the influence of vildagliptin on model-assessed -cell function in patients with type 2 diabetes and mild hyperglycemia. J Clin Endocrinol Metab. 2008 Jan;93(1):103-9. doi: 10.1210/jc.2007-1639. Epub 2007 Oct 9. PMID 17925336